CLINICAL TRIAL: NCT04607161
Title: External Validation of Two Prediction Models for Adequate Bowel Preparation in Asia: A Prospective Study
Brief Title: External Validation of Models for Predicting Inadequate Bowel Preparation
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IBPV-V1.0
Record Dates: First submitted 2020-10-25; First posted 2020-10-29 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Colonoscopy; Predictive Model; External Validation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
In order to obtain the risk level of patients with intestinal insufficiency through simple indicators, many foreign scholars have studied and developed their own prediction models. However, the current guideline indicates that there is insufficient evidence to recommend the use of a specialized predictive model for clinical practice.There are few studies on external validation of existing prediction models.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing colonoscopy.
* patients older than 18 years.

Exclusion Criteria:

* Emergency colonoscopy.
* Have a serious medical condition, such as heart failure, acute liver failure, severe kidney disease (dialysis or predialysis patients) or New York heart association class iii-iv.
* Pregnant or breastfeeding.
* No bowel preparation or poor compliance (no bowel preparation as instructed or laxatives < 90% of prescribed dose).
* Refuse to sign informed consent.
* The patient was rescheduled after the previous colonoscopy due to insufficient bowel preparation.
* Temporarily change to colonoscopy for other reasons.
* Incomplete colonoscopy due to insufficient parenteral preparation.
* Lack of complete data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
discrimination | cross-sectional analyses in 2020
  Compare the area under the curve (AUC) between predictive models and acutal bowel preparation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China

REFERENCES:
- [Derived] Yuan X, Gao H, Liu C, Wang W, Xie J, Zhang Z, Xu L. External validation of two prediction models for adequate bowel preparation in Asia: a prospective study. Int J Colorectal Dis. 2022 Jun;37(6):1223-1229. doi: 10.1007/s00384-022-04156-0. Epub 2022 Apr 25. PMID 35467123